CLINICAL TRIAL: NCT04018573
Title: Developing an HIV Prevention Intervention for Young MSM Through Improved Parent-child Communication
Brief Title: Testing an Online Intervention to Improve Parents' Communication With Gay and Bisexual Sons About Sex and HIV
Acronym: PATHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Huebner, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MH112445; R34MH112445 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-07-12 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Support Film (Active Comparator): Parents will watch Lead with Love, a 35-minute documentary style film designed to provide support, information, and behavioral guidance to parents with a lesbian, gay, or bisexual child. One month later, parents will look over material that reviews the major points of the film. All of this material is presented online via our webapp.
  Interventions: Behavioral: Parent Support Film
- Parent Support Film + PATHS Sexual Communication Toolkit (Experimental): Parents in this arm will have the option of watching Lead with Love, and then will engage with our parent toolkit, designed to increase the frequency and quality of parent-child communication about HIV and condoms. One month later, parents will engage with booster content, customized to address their self-reported barriers to communicating with their sons. All of this material is presented online via our webapp.
  Interventions: Behavioral: PATHS Sexual Communication Toolkit; Behavioral: Parent Support Film

INTERVENTIONS:
Behavioral: PATHS Sexual Communication Toolkit — The PATHS Sexual Communication Toolkit is a self-guided, online intervention. The toolkit is comprised of 6 modules, covering a range of topics relevant to increasing parents' motivation, self-efficacy, and intention for communicating about sex. Material is presented in a variety of modalities (e.g., text, videos of experts, videos of other parents describing their experiences). Parents set personalized goals for themselves regarding activities and conversations they want to have with their sons, selecting from a menu of options provided by the intervention. A 1-month booster module queries parents about whether they have achieved their goals, and provides customized content to support the behaviors parents have yet to enact.
  Arms: Parent Support Film + PATHS Sexual Communication Toolkit
Behavioral: Parent Support Film — Lead with Love is a 35-minute "education entertainment" film created to provide support, information, and behavioral guidance to parents of lesbian, gay, or bisexual (LGB) children. Drawing from stage-based models of behavior change, and social cognitive theory, it aims to help parents progress through the process of coming to accept their child's sexual orientation, recognizing the importance of their behaviors and reactions to their child's health, and accepting their child's sexual orientation, and engaging in behaviors that are more supportive and less rejecting. This is achieved by telling the true stories of four families and how they responded to the news that their child was LGB, and by having experts (psychologists, teachers, clergy) provide information and guidance.
  Other Names: Lead with Love

SUMMARY:
Young men who have sex with men (MSM) are at high risk for HIV infection in the United States, representing 80% of all infections among youth ages 14-24, and 92% of infections among boys ages 14-19. Despite these risks, the field has not even one HIV prevention intervention shown to be effective in decreasing sexual risks or increasing HIV testing among adolescent MSM (AMSM). Historically, reaching AMSM for HIV prevention has been challenging, given their relative geographic isolation and lack of access to traditional gay congregating spaces (e.g., bars and many gay-related social networking websites). However, the investigators have developed a novel online platform for delivering interventions to parents of LGB youth that currently sees thousands of visitors each year. HIV prevention advocates have identified parents of AMSM as an untapped resource for reducing HIV risk in this population. Parent-child communication about sex has well-demonstrated associations with adolescent risk behaviors, and interventions with parents of heterosexual youth have been shown to be effective in increasing parent-adolescent communication, and thereby, reducing adolescent health risks. Thus, the aim of the proposed study is to pilot test the efficacy of an online intervention to increase and improve parent communication with AMSM about sexuality and HIV, with the ultimate goal of decreasing adolescent sexual risk and increasing HIV testing. This will be achieved by randomizing parents who come to seek resources on the investigators' existing website to receive either (a) a film designed to support parents of LGB youth, or (b) that film + the online communication intervention materials, and then gathering longitudinal, online data from parents in both study arms and their AMSM sons over a 2-4 month period. It is hypothesized that parents in the intervention group will increase their communication with their sons about HIV and condoms.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child with all of the following characteristics:

  1. cisgender male
  2. age 14-22
  3. self-identify as gay or bisexual
  4. lives in the same house with parent at least 2 days per week.

     Exclusion Criteria:
* Child with known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Health Communication Checklist score -- Parents | Parents are queried about whether they engaged in these behaviors at three time points: baseline, 4-6 week follow-up, and 8-12 week follow-up. We will assess change from baseline to each of the two followup points.
  This is a new measure developed for this pilot study. Thus, we will first examine the measure's reliability and validity. Assuming acceptable psychometric properties, this will be the primary outcome measure. The checklist queries parents and children whether they have engaged in four different activities specifically recommended by our intervention: providing information about HIV, providing information about correct condom usage, providing information about condom acquisition, and supporting HIV testing. For each of those four activities, families have multiple ways to do the activity (e.g., for providing information about correct condom use, parents can: send a video, explain the process, or demonstrate the process). Thus, the checklist queries 11 specific behaviors. Families are coded as having completed the activity if they have engaged in any one of the multiple behaviors congruent with the corresponding activity. Thus, scores on the measure range from 0-4.
Change in Sexual Health Communication Checklist score -- Child | Sons are queried about whether their parents engaged in these behaviors at baseline and at 12 week followup. We will assess change from baseline to followup.
  This is a new measure developed for this pilot study. Thus, we will first examine the measure's reliability and validity. Assuming acceptable psychometric properties, this will be the primary outcome measure. The checklist queries parents and children whether they have engaged in four different activities specifically recommended by our intervention: providing information about HIV, providing information about correct condom usage, providing information about condom acquisition, and supporting HIV testing. For each of those four activities, families have multiple ways to do the activity (e.g., for providing information about correct condom use, parents can: send a video, explain the process, or demonstrate the process). Thus, the checklist queries 11 specific behaviors. Families are coded as having completed the activity if they have engaged in any one of the multiple behaviors congruent with the corresponding activity. Thus, scores on the measure range from 0-4.

SECONDARY OUTCOMES:
Change in parent intentions for sexual health communication | Parents are given this measure at baseline, immediately post-intervention, and at 4-6 week follow-up after engaging with booster material. We will assess change from baseline to post intervention and from baseline to 4-6 week followup.
  This is a new measure developed for this pilot study. It assesses parents' intentions in the "next several weeks" to engage in 11 specific sexual health activities with their sons (e.g., demonstrating condom use, taking son to get tested for HIV).
Change in Parent-Adolescent Sexual Health Communication Assessment | Parents are queried at baseline, 8-week followup, and 12-week followup. Sons are queried at baseline and 12-week followup.
  This measure contains subscales assessing: (a) sexual health communication frequency, (b) sexual health communication quality, and (c) negative emotionality during sexual health communication. There are both parent and child reports.
Change in condom-use self efficacy | For parents: change from baseline to immediate post-intervention. For sons: change from baseline to 12-week follow-up
  11-item scale assessing participants' confidence in their ability to correctly use and acquire condoms. Assessed in parents and sons.

OTHER OUTCOMES:
Change in HIV knowledge | For parents: change from baseline to immediate post-intervention. For sons: change from baseline to 12-week follow-up.
  17-item true/false scale assessing factual knowledge about HIV
Change in condom knowledge | For parents: change from baseline to immediate post-intervention. For sons: change from baseline to 12-week follow-up
  Participants are presented with 13 statements, and are asked to identify which 6 describe accurate steps in correct condom use.
Change in self-efficacy for communicating with a child about condoms | Change from baseline to (a) immediate post-intervention, (b) 8 week followup, and (c) 12 week followup.
  6-items assessing parents' confidence in their ability to talk with their sons about condom use
Change in outcome expectancy for condom communication | Change from baseline to (a) immediate post-intervention, (b) 8 week followup, and (c) 12 week followup.
  12-item scale assessing the degree to which parents believe positive or negative things would happen if they talked to their son about condoms.

CONTACTS AND LOCATIONS:
Overall Officials: David M Huebner, PhD, MPH, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Huebner DM, Barnett AP, Baucom BRW, Guilamo-Ramos V. Effects of a Parent-Focused HIV Prevention Intervention for Young Men Who have Sex with Men: A Pilot Randomized Clinical Trial. AIDS Behav. 2023 May;27(5):1502-1513. doi: 10.1007/s10461-022-03885-1. Epub 2022 Nov 10. PMID 36352294